CLINICAL TRIAL: NCT04499066
Title: Peripartum Mental Health Cohort Study in Guangzhou
Status: Recruiting | Type: Observational
Sponsor: Guangzhou Women and Children's Medical Center (Other)
Responsible Party: Principal Investigator, Xiu Qiu, Director of the Born in Guangzhou Cohort Study, Guangzhou Women and Children's Medical Center
Other Study IDs: 2018053101
Record Dates: First submitted 2020-07-21; First posted 2020-08-05 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Depression; Anxiety
Keywords: Peripartum; Mental health; Risk factors; Pregnancy outcome; Cohort
MeSH Terms: conditions — Depression; Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — During pregnancy: maternal blood, urine and stool. At delivery: cord, cord blood and placenta. During infancy: dry blood spot and blood of children.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to determine the incidence,development trajectory and risk factors of the main peripartum mental health problems as well as explore its adverse outcomes.

DETAILED DESCRIPTION:
Peripartum mental health problems (such as anxiety and depression), affecting more than 20% of mothers, is one of the most common complications around childbirth and gradually have become global public health issues. However, little is known about the course of peripartum mental health problems and possible fluctuations, as well as related risk factors among Chinese women. In addition, there are no effective prediction and preventive strategies for postpartum depression. The Peripartum Mental Health Cohort Study in Guangzhou will collect the epidemiological, clinical information and biological specimens across pregnancy and childbirth to establish trajectory of peripartum mental health and identify the factors influencing the fluctuations and build a comprehensive prediction model of postpartum depression, as well as explore its adverse outcomes. This study would help to determine the timing of screening and target interventions to improve women's and their offspring's health.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women with <20 weeks of gestation
2. Pregnant women intended to eventually deliver in Guangzhou Women and Children's Medical Center
3. Permanent residents or families intended to remain in Guangzhou with their child for more than 3 years

Exclusion Criteria:

1. Combined with heart disease, hypertension, diabetes or hyperthyroidism
2. Taking anti-depressants and other treatments for depression
3. Participants was in infection status when the biological samples were collected

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women before 20 weeks of gestation
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2012-02-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2038-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of prevalence of maternal prenatal depression | before 20th gestational week, after 33th gestational week and prior to delivery
  Using Self-rating Depression Scale (SDS) to assess maternal depressive symptoms during pregnancy. SDS scores ≥53 is defined as prenatal depressive symptoms.
Change of prevalence of maternal postpartum depression in the first year after delivery | 6 weeks, 6 months and 1 year after delivery
  Using Edinburgh Postnatal Depression Scale (EPDS) to assess postpartum depressive symptoms. EPDS scores ≥13 is defined as postpartum depressive symptoms.

SECONDARY OUTCOMES:
Change of prevalence of maternal anxiety during pregnancy | before 20th gestational week, after 33th gestational week and prior to delivery
  Using Self-rating Anxiety Scale (SAS) to assess maternal anxiety during pregnancy. SAS scores ≥50 is defined as anxiety.
Level of maternal cortisol during pregnancy | During period of 2-3 trimesters of pregnancy
  Using women's blood samples to test the concentration of cortisol.
Levels of maternal inflammatory factors during pregnancy | During period of 2-3 trimesters of pregnancy
  Using women's blood samples to test the concentration of inflammatory factors, including CRP, IL-6, TNF-α, etc.
Prevalence of preterm birth, small for gestational age, low birth weight | At delivery
  Obtained from electronic medical records.
Child's neurodevelopment at early childhood | At child's age of 1 year
  Assessed by using the Gesell Developmental Schedules, which includes adaptive, gross motor, fine motor, language, and social function domains. Higher score in each domain is considered a better outcome, while no more than 85 is defined as suspected development delay.

CONTACTS AND LOCATIONS:
Overall Officials: Xiu Qiu, PhD, Principal Investigator — Guangzhou Women and Children's Medical Center
Locations (1):
- Guangzhou Women and Children's Medical Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Qiu X, Lu JH, He JR, Lam KH, Shen SY, Guo Y, Kuang YS, Yuan MY, Qiu L, Chen NN, Lu MS, Li WD, Xing YF, Zhou FJ, Bartington S, Cheng KK, Xia HM. The Born in Guangzhou Cohort Study (BIGCS). Eur J Epidemiol. 2017 Apr;32(4):337-346. doi: 10.1007/s10654-017-0239-x. Epub 2017 Mar 20. PMID 28321694